CLINICAL TRIAL: NCT05094986
Title: Pilot of a Complex Intervention to Improve Initial Medication Adherence to Cardiovascular and Diabetes Treatments in Primary Care
Brief Title: Feasibility and Acceptability of a Complex Intervention to Improve Initial Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Parc Sanitari Sant Joan de Déu (Other); Institut Català de la Salut (Other); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other); Col·legi de Farmacèutics de la Província de Barcelona (Other); CIBER of Epidemiology and Public Health (Unknown)
Responsible Party: Principal Investigator, Maria Rubio-Valera, Head of Quality and Patient Safety, Fundació Sant Joan de Déu
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19/198-P
Record Dates: First submitted 2021-10-08; First posted 2021-10-26 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Adherence, Medication
Keywords: Pilot Study; Feasibility Study; Complex Intervention; Real-World Data; Cardiovascular Disease; Diabetes Mellitus
MeSH Terms: conditions — Medication Adherence; Cardiovascular Diseases; Diabetes Mellitus | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Masking Description: PC patients: Patients from the intervention PCCs received the IMA intervention but were not aware of the group they were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: IMA Intervention (Experimental): General practitioners (GP) applied the IMA intervention to all patients receiving a new prescription for pharmacological treatments of cardiovascular disease or diabetes.
  Following the IMA intervention, nurses and community pharmacists offered information support in line with the information provided by the GP. Professionals had the intervention support tools available (leaflets, website and dispensing alert in community pharmacies).
  Interventions: Behavioral: Initial Medication Adherence (IMA) Intervention
- Control group (Active Comparator): Healthcare professionals from the control group prescribed medication and provided information as usual.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Initial Medication Adherence (IMA) Intervention — The IMA intervention promotes health literacy and patient participation in the decision-making process during the recommendation and prescription of a new drug for the management of cardiovascular disease and diabetes. The IMA intervention has four main components: 1. Training for healthcare professionals (GPs, nurses, and community pharmacists) on non-initiation, shared-decision making, health literacy and use of decision aids; 2. Intervention support tools; decision aids (leaflets and website) and implementation tools (dispensing alert in community pharmacies when dispensing insulins and antiplatelet drugs); 3. Shared decision-making process during the GP's consultation; and 4. Information support provided by the nurses and community pharmacists that use the intervention decision aids to explore the patients' doubts and standardise the discourse between primary healthcare professionals.
  Arms: Intervention group: IMA Intervention
Other: Usual Care — Patients received the usual care when being prescribed a new prescription for treatments of cardiovascular disease or diabetes. Nurses and community pharmacists were asked to also provide usual care to those patients. Community pharmacists from the control group had the dispensing alert available when dispensing insulins and antiplatelet drugs.
  Arms: Control group

SUMMARY:
This pilot study aims to test the feasibility of the following effectiveness and cost-effectiveness evaluation using Real-World Data.

DETAILED DESCRIPTION:
A cluster non-randomised pilot study with an embedded process evaluation was carried out to test the feasibility of the definitive cluster randomised controlled trial (cRCT). The cRCT will aim to evaluate the effectiveness and cost-effectiveness of the Initial Medication Adherence (IMA) intervention in comparison to usual care, to increase initiation of pharmacological treatments for CVD and diabetes (antihypertensive drugs, hypolipidemic drugs, antiplatelet drugs, and insulin and oral antidiabetics) prescribed in Primary Care (PC).

The pilot study was conducted in five PC centres (PCC) in Catalonia (Spain), two were assigned to the control group and three to the intervention group. There were two target participants, the implementation targeted professionals (general practitioners (GP), nurses, and community pharmacists), and the population targeted by the intervention, PC patients.

The IMA intervention provided healthcare professionals with the knowledge, skills, and tools to help the patient make an informed and shared decision with the GP to initiate a new CVD or diabetes treatment. Professionals were trained on the problem of non-initiation, communication skills, health literacy, and the use of decision aids (leaflets, website).

ELIGIBILITY:
Inclusion Criteria:

Primary healthcare professionals and pharmacists who:

• Agree to participate in the pilot study.

Primary care patients who:

* Are prescribed a new treatment of cardiovascular disease o diabetes by a GP who participates in the clinical trial.
* Are >18 years old.
* Do not reject to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of clinical registries related to diabetes mellitus II | 5 months before and after recruitment
  Rate of registries recorded five months before and after the prescription of:
  * Glycated haemoglobin
  * Glomerular filtrate
  * Blood glucose
Rate of clinical registries related to dyslipidemia | 5 months before and after recruitment
  Rate of registries recorded five months before and after the prescription of:
  * Total colesterol
  * HDL cholesterol
  * LDL colesterol
Rate of clinical registries related to hypertension | 2 months before and after recruitment
  Rate of registries recorded one to two months before and after the prescription of:
  * Systolic blood pressure
  * Diastolic blood pressure
Rate of clinical registries related to cardiovascular risk | 5 months before and after recruitment
  Rate of registries recorded five months before and after the prescription of:
  • REGICOR
Rate of use of services | 5 months before and after recruitment
  Rate of use of services recorded five months before and after the prescription of:
  * Visits to primary care (nurse, GP)
  * Referrals to secondary care
  * Productivity losses (sick leave days)
  * Outpatient diagnostic tests

SECONDARY OUTCOMES:
Active diagnosis registry | 5 months before and after recruitment
  Proportion of patients with a new prescription of cardiovascular disease and diabetes treatments and an active diagnosis in the electronic system.
Missing registries | 5 months before and after recruitment
  Number of registries missing.
Outliers registries | 5 months before and after recruitment
  Number of registries with values out of their range.

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - CAP Cornellà de Llobregat (La Gavarra), Cornellà de Llobregat, Barcelona
  - Centro de Asistencia Primaria (CAP) Dr. Pujol i Capsada (CAP Pujol i Capsada), el Prat de Llobregat, Barcelona
  - CAP Dr. Bartomeu Fabrés Anglada Gava 2, Gavà, Barcelona
  - CAP Florida Nord (CAP la Florida), L'Hospitalet de Llobregat, Barcelona
  - CAP Florida Sud (CAP la Florida), L'Hospitalet de Llobregat, Barcelona

IPD SHARING:
Plan to Share IPD: No
The research team is not the data owner as they are only re-using information that is the property of the public health institutions in Catalonia.
  Consequently, meta-data cannot be published by the authors nor data can be identified with a DOI.

REFERENCES:
- [Derived] Corral-Partearroyo C, Sanchez-Vinas A, Gil-Girbau M, Penarrubia-Maria MT, Aznar-Lou I, Serrano-Blanco A, Carbonell-Duacastella C, Gallardo-Gonzalez C, Olmos-Palenzuela MDC, Rubio-Valera M. Improving Initial Medication Adherence to cardiovascular disease and diabetes treatments in primary care: Pilot trial of a complex intervention. Front Public Health. 2022 Dec 6;10:1038138. doi: 10.3389/fpubh.2022.1038138. eCollection 2022. PMID 36561857